CLINICAL TRIAL: NCT02437279
Title: Feasibility Study to Identify the Optimal Adjuvant Combination Scheme of Ipilimumab and Nivolumab in Stage III Melanoma Patients
Brief Title: Study to Identify the Optimal Adjuvant Combination Scheme of Ipilimumab and Nivolumab in Melanoma Patients
Acronym: OpACIN
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N14OPC; CA209-278 (Other Grant/Funding Number: BMS); NL51280.031.14 (Registry Identifier: CCMO register)
Record Dates: First submitted 2015-04-13; First posted 2015-05-07 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Stage III Skin Melanoma
Keywords: Palpable; Stage III; Skin melanoma; Ipilimumab; Nivolumab; Surgery
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Post-surgery infusion for 12 weeks with the combination of ipilimumab+nivolumab
  Interventions: Procedure: Surgery of the tumor; Drug: Infusion with ipilimumab 3 mg/kg q3wks; Drug: Infusion with nivolumab 1 mg/kg q3wks
- Arm B (Active Comparator): A split design 6 weeks upfront surgery and 6 weeks post-surgery infusion with the combination of ipilimumab+nivolumab
  Interventions: Procedure: Surgery of the tumor; Drug: Infusion with ipilimumab 3 mg/kg q3wks; Drug: Infusion with nivolumab 1 mg/kg q3wks

INTERVENTIONS:
Procedure: Surgery of the tumor
Drug: Infusion with ipilimumab 3 mg/kg q3wks
Drug: Infusion with nivolumab 1 mg/kg q3wks

SUMMARY:
This is a two-arm Phase 1b feasibility trial consisting of 20 patients receiving the combination of ipilimumab+nivolumab, either adjuvant, or split neo-adjuvant and adjuvant.

DETAILED DESCRIPTION:
Patients with stage III melanoma with palpable disease, naïve for CTLA-4/PD-1/PD-L1 immunotherapy, will be treated either post-surgery for 12 weeks with the combination of ipilimumab+nivolumab or in a split design for 6 weeks upfront surgery and for 6 weeks postsurgery. It is a two-arm Phase 1b feasibility trial consisting of 20 patients, 10 in each arm.

At different timepoints tumor biopsies and blood for PBMCs will be taken for translational research. Also scans will be done on specific timepoints.

The study will be held to determine safety, feasibility, and the immune-activating capacity of short-term combined neo-adjuvant and adjuvant ipilimumab + nivolumab. And to determine relapse free survival (RFS), any late adverse events, pharmacokinetics/pharmacodynamics, and the correlation between RFS and changes in neo-antigen specific T cell response.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* World Health Organization (WHO) Performance Status 0 or 1
* Histologically confirmed stage IIIB metastatic cutaneous melanoma, palpable disease (non-transit only) of the axilla or groin
* Patient willing to undergo triple tumor biopsies during screening and in case of disease progression
* No prior immunotherapy targeting CTLA-4, PD-1 or PD-L1
* No immunosuppressive medications within 6 months prior study inclusion
* Presence of at least two of the defined HLA alleles (Table 1, see appendix)
* Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Neutrophils

  ≥1.5x109/L, Platelets ≥100 x109/L, Hemoglobin ≥5.5 mmol/L, Creatinine ≤1.5x ULN, AST ≤1.5 x ULN, ALT ≤ 1.5 x ULN, Bilirubin ≤1.5 X ULN
* normal LDH
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of ipilimumab+nivolumab
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product
* Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception

Exclusion Criteria:

* Distantly metastasized melanoma
* Subjects with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for subjects with vitiligo or resolved childhood asthma/atopy
* Prior CTLA-4 or PD-1/PD-L1 targeting immunotherapy
* Radiotherapy prior or post surgery within this trial
* Patients will be excluded if they are positive test for hepatitis B virus surface antigen (HBVsAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Patients will be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Allergies and Adverse Drug Reaction

  * History of allergy to study drug components
  * History of severe hypersensitivity reaction to any monoclonal antibody
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events;
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids;
* Use of other investigational drugs before study drug administration 30 days and 5 half-times before study inclusion
* Pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-24 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The alteration in magnitude of the neo-antigen specific T cell response in the time interval pre- to post-adjuvant therapy in peripheral blood | 12 weeks from baseline
  To this purpose the immunogenic mutational load of each patient's melanoma will be determined by DNA and RNA sequencing from baseline biopsies (3x14g, 5ug tumor DNA). Proteasomal degradation and peptide presentation in HLA will be predicted in silico. MHC-tetramer staining containing the predicted peptides will be done as described before [2]. In addition, the effect of therapy on intratumoral T cell responses to obtain better insight into the mode of action of therapy will be analyzed. Identified neo-antigen specific T cells will be analyzed with respect to their phenotype and immunologic function (intracellular cytokine staining, lytic function as determined by CD107 staining, and coculture with APC presenting the cognate antigen).
Safety as measured by SUSARs. | 12 weeks from baseline
The alteration in breadth of the neo-antigen specific T cell response in the time interval pre- to post-adjuvant therapy in peripheral blood | 12 weeks from baseline
  To this purpose the immunogenic mutational load of each patient's melanoma will be determined by DNA and RNA sequencing from baseline biopsies (3x14g, 5ug tumor DNA). Proteasomal degradation and peptide presentation in HLA will be predicted in silico. MHC-tetramer staining containing the predicted peptides will be done as described before [2]. In addition, the effect of therapy on intratumoral T cell responses to obtain better insight into the mode of action of therapy will be analyzed. Identified neo-antigen specific T cells will be analyzed with respect to their phenotype and immunologic function (intracellular cytokine staining, lytic function as determined by CD107 staining, and coculture with APC presenting the cognate antigen).
Feasibility as measured adherence to the timelines in the study protocol. | 12 weeks from baseline

SECONDARY OUTCOMES:
Recurrence Free Survival, as determined according to RECIST 1.1 criteria. | Until progression, median 10 months.
Rate of adverse events and late adverse events | Until end of follow-up, median 3 years.
Type of adverse events and late adverse events | Until end of follow-up, median 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Blank, MD PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Zijlker LP, van der Burg SJC, Blank CU, Zuur CL, Klop WMC, Wouters MWMJ, van Houdt WJ, van Akkooi ACJ. Surgical outcomes of lymph node dissections for stage III melanoma after neoadjuvant systemic therapy are not inferior to upfront surgery. Eur J Cancer. 2023 May;185:131-138. doi: 10.1016/j.ejca.2023.03.003. Epub 2023 Mar 7. PMID 36989829
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215
- [Derived] Versluis JM, Reijers ILM, Rozeman EA, Menzies AM, van Akkooi ACJ, Wouters MW, Ch'ng S, Saw RPM, Scolyer RA, van de Wiel BA, Schilling B, Long GV, Blank CU. Neoadjuvant ipilimumab plus nivolumab in synchronous clinical stage III melanoma. Eur J Cancer. 2021 May;148:51-57. doi: 10.1016/j.ejca.2021.02.012. Epub 2021 Mar 15. PMID 33735809
- [Derived] Rozeman EA, Hoefsmit EP, Reijers ILM, Saw RPM, Versluis JM, Krijgsman O, Dimitriadis P, Sikorska K, van de Wiel BA, Eriksson H, Gonzalez M, Torres Acosta A, Grijpink-Ongering LG, Shannon K, Haanen JBAG, Stretch J, Ch'ng S, Nieweg OE, Mallo HA, Adriaansz S, Kerkhoven RM, Cornelissen S, Broeks A, Klop WMC, Zuur CL, van Houdt WJ, Peeper DS, Spillane AJ, van Akkooi ACJ, Scolyer RA, Schumacher TNM, Menzies AM, Long GV, Blank CU. Survival and biomarker analyses from the OpACIN-neo and OpACIN neoadjuvant immunotherapy trials in stage III melanoma. Nat Med. 2021 Feb;27(2):256-263. doi: 10.1038/s41591-020-01211-7. Epub 2021 Feb 8. PMID 33558721